CLINICAL TRIAL: NCT02675101
Title: Nuts and Olestra for Persistent Organic Pollutant Reduction (NO-POPs) Trial: A Pilot Investigation
Brief Title: Nuts and Olestra for Persistent Organic Pollutant Reduction (NO-POPs) Trial
Acronym: NO-POPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Jose R Suarez, MPH, MD, PhD, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160096
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Persistent Organic Pollutants; Endocrine Disrupting Chemicals; Endocrine Disruptor Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whole nuts (Active Comparator): Participants will be advised on maintaining an iso-caloric diet by a Registered Dietitian. During the 6-month intervention, study subjects will consume a combination of whole almonds and walnut pieces, a total of 110 g per day. Participants will pick up supplies and be weighed 1-2 times per month for six months. Participants will also maintain a diary of their intake using an automated system. Walnuts and almonds will be provided to participants for the duration of the study.
  Interventions: Other: Whole Nuts
- Olestra: Fat Free Pringles (Experimental): Participants will be advised on maintaining an iso-caloric diet by a Registered Dietitian. During the 6-month intervention, study subjects will consume 29 potato crisps per day, which is approximately 18 g olestra/day. Participants will pick up supplies and be weighed 1-2 times per month for six months. Participants will also maintain a diary of their intake using an automated system. Fat free Pringles will be provided to participants for the duration of the study.
  Interventions: Other: Olestra: Fat Free Pringles
- Vegetable Oil: Original Pringles (Placebo Comparator): Participants will be advised on maintaining an iso-caloric diet by a Registered Dietitian. During the 6-month intervention, study subjects will consume 29 potato crisps per day, which is approximately 17.4 g oil/day. Participants will pick up supplies and be weighed 1-2 times per month for six months. Participants will also maintain a diary of their intake using an automated system. Original Pringles will be provided to participants for the duration of the study.
  Interventions: Other: Vegetable Oil: Original Pringles

INTERVENTIONS:
Other: Whole Nuts — Participants will be advised on maintaining an iso-caloric diet. Aside consuming nuts, the remaining composition of the prescribed diet will be based on individual preferences. During the 6-month intervention, study subjects will meet with study staff every 2-3 weeks to weigh in, pick up food supplies and complete a questionnaire on compliance. All participants will have contact with the project coordinator/study dietitian a minimum of every 1-2 weeks either in-person, telephone, email and text message contacts for support, behavioral guidance and strategies. Both walnuts and almonds will be provided to participants in the whole nut study arm.
  Arms: Whole nuts
Other: Olestra: Fat Free Pringles — Participants will be advised on maintaining an iso-caloric diet. Aside consuming fat free potato crisps, the remaining composition of the prescribed diet will be based on individual preferences. During the 6-month intervention, study subjects will meet with study staff every 2-3 weeks to weigh in, pick up food supplies and complete a questionnaire on compliance. All participants will have contact with the project coordinator/study dietitian a minimum of every 1-2 weeks either in-person, telephone, email and text message contacts for support, behavioral guidance and strategies. Fat Free Pringles will be provided to participants in the olestra study arm.
  Arms: Olestra: Fat Free Pringles
Other: Vegetable Oil: Original Pringles — Participants will be advised on maintaining an iso-caloric diet. Aside consuming potato crisps, the remaining composition of the prescribed diet will be based on individual preferences. During the 6-month intervention, study subjects will meet with study staff every 2-3 weeks to weigh in, pick up food supplies and complete a questionnaire on compliance. All participants will have contact with the project coordinator/study dietitian a minimum of every 1-2 weeks either in-person, telephone, email and text message contacts for support, behavioral guidance and strategies. Original Pringles will be provided to participants in the vegetable oil study arm.
  Arms: Vegetable Oil: Original Pringles

SUMMARY:
Persistent organic pollutants (POPs) are mostly fat-soluble halogenated chemicals with very long half-lives. POPs are endocrine disruptors, associated with increased risk for diabetes, alterations in thyroid function, and cardiovascular disease in humans. POPs concentrations increase with age because of their persistence, bioaccumulation and poor excretion. The almost ubiquitous presence of endocrine disrupting POPs in US adults is a substantial public health concern, particularly because there is no established treatment to reduce body concentrations of POPs. Most POPs are excreted in bile due to their lipophilic nature. However, a substantial amount is reabsorbed in the small intestine and returns to the blood stream (entero-hepatic circulation). The objective of this pilot study is to conduct a 6-month randomized controlled trial of Nuts and Olestra to enhance the excretion of POPs among 45 healthy adults aged 45 to 70 years with BMIs between 18-30 kg/m2. This study has 3 treatment arms: A) Whole nuts with high fat content (almonds and walnuts; 110g total/day, n=15), B) Olestra: Fat Free PringlesTM potato chips (≈29 crisps, 18g of Olestra/day; n=15), C) Vegetable oil: Original PringlesTM potato chips (≈29 crisps, 17.4g of oil/day; n=15). The investigators aim to measure change in concentrations of 24 POPs in feces after 4 days of treatment and in blood at 6 months.

DETAILED DESCRIPTION:
Persistent organic pollutants (POPs) are mostly fat-soluble halogenated chemicals with very long half-lives. POPs are endocrine disruptors, and have been associated with increased risk for diabetes, alterations in thyroid function, hypertension, dyslipidemia and neurobehavioral alterations in studies of children, and adults including the elderly. Some of the most prevalent POPs include organochlorine pesticides, polychlorinated biphenyls (PCBs) and polybrominated diphenyl ethers (PBDEs).

Most POPs are excreted in bile due to their lipophilic nature. However, a substantial amount is reabsorbed in the small intestine and returns to the blood stream (entero-hepatic circulation). Two small clinical trials found that bile acid sequestrants (cholestyramine, cholestimide) enhanced the fecal excretion of organochlorines after 2-3 days of treatment and significantly lowered their blood concentrations at 6 months. One pilot trial reported decreases in blood PCB concentrations in adults after a 1 year treatment with fat-free potato crisps made with olestra, a non-absorbable synthetic fat, versus standard potato crisps. POPs were thought to bind to olestra and be excreted in the feces. Replication of this finding is needed. Nuts, could yield similar effects. Nuts are foods with high-fat content which are incompletely absorbed in the intestine (21-24% of calorie not absorbed).

As people age, the body burdens of POPs increase. The almost ubiquitous presence of endocrine disrupting POPs in US adults is a substantial public health concern, particularly because there is no established treatment to reduce body concentrations of POPs. There is potential for dietary interventions to have an important role in the reduction of POPs at a population level due to their and low cost and wide use.

The investigators aim to measure 24 POPs (9 OC pesticides, 10 PCBs, 5 PBDEs) in blood (all participants) and in stool samples (only in a subset of 10 participants per treatment arm) before and during the treatment period. The specific aims of this pilot study are to:

1. Assess the effectiveness of recruitment strategies, acceptance and compliance of the treatment arms, and establishing the feasibility of conducting a larger trial.
2. Conduct preliminary testing of the hypotheses: Consumption of olestra (fat free Pringles): A) increases the fecal content (excretion) of POPs, and B) decreases blood levels of POPs, compared to the control arm (standard crisps).
3. Conduct preliminary testing of the hypotheses: Consumption of nuts: A) increases the fecal content (excretion) of POPs, and B) decreases blood levels of POPs, compared to the control arm (standard crisps).

ELIGIBILITY:
Inclusion Criteria:

* Reside in the San Diego area
* BMI ≥18.0 kg/m2 and ≤30 kg/m2
* Non-smoker
* Willing and able to participate in clinic visits, bi-monthly supply pick-up, telephone and Internet communications at specified intervals
* Able to provide data through questionnaires and by telephone
* Willing to maintain contact with the investigators for 6 months
* Willing to allow blood collections
* Willing to provide stool samples
* No known allergy to tree nuts
* No digestive issues with olestra, chips, or nuts

Exclusion Criteria:

* Nut allergies
* Smoker
* Diabetes, kidney disease or liver disease
* Concurrent acute or chronic gastro-intestinal conditions (e.g. inflammatory bowel disease, irritable bowel syndrome, concurrent diarrhea from any cause)
* Familial hypercholesterolemia
* Clotting problems or use of Coumadin,
* Inability to participate in physical activity because of severe disability
* History or presence of a co-morbid diseases for which diet modification may be contraindicated
* Self-reported pregnancy or breastfeeding or planning a pregnancy within the next year
* Currently actively involved in another diet intervention study or a weight loss program
* A history or presence of a significant psychiatric disorder or any other condition that, in the investigator's judgement, would interfere with participation in the trial

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in blood levels of persistent organic pollutants (POPS) in response to being assigned an olestra -enriched diet (fat-free Pringles) compared to a diet enriched with vegetable oil (original Pringles) over a 6-month period | 6 months
Change in fecal excretion of persistent organic pollutants (POPS) in response to being assigned an olestra -enriched diet (fat-free Pringles) compared to a diet enriched with vegetable oil (original Pringles) over a 6-month period | 6 months

SECONDARY OUTCOMES:
Change in blood levels of persistent organic pollutants (POPS) in response to being assigned a nut-enriched diet compared to a diet enriched with vegetable oil (original Pringles) over a 6-month period | 6 months
Change in fecal excretion of persistent organic pollutants (POPS) in response to being assigned a nut-enriched diet compared to a diet enriched with vegetable oil (original Pringles) over a 6-month period | 6 months

OTHER OUTCOMES:
Change in blood lipids in response to being assigned an olestra -enriched diet (fat-free Pringles), a vegetable oil-enriched diet (original Pringles) or a nut-enriched diet over a 6-month period, as an exploratory aim. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Suarez, MPH, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Contreras Lopez MC. Determination of potentially bioaccumulating complex mixtures of organochlorine compounds in wastewater: a review. Environ Int. 2003 Mar;28(8):751-9. doi: 10.1016/S0160-4120(02)00120-4. PMID 12605924
- [Background] Hinck JE, Norstrom RJ, Orazio CE, Schmitt CJ, Tillitt DE. Persistence of organochlorine chemical residues in fish from the Tombigbee River (Alabama, USA): Continuing risk to wildlife from a former DDT manufacturing facility. Environ Pollut. 2009 Feb;157(2):582-91. doi: 10.1016/j.envpol.2008.08.021. Epub 2008 Oct 11. PMID 18851891
- [Background] Dougherty CP, Henricks Holtz S, Reinert JC, Panyacosit L, Axelrad DA, Woodruff TJ. Dietary exposures to food contaminants across the United States. Environ Res. 2000 Oct;84(2):170-85. doi: 10.1006/enrs.2000.4027. PMID 11068931
- [Background] Schafer KS, Kegley SE. Persistent toxic chemicals in the US food supply. J Epidemiol Community Health. 2002 Nov;56(11):813-7. doi: 10.1136/jech.56.11.813. PMID 12388566
- [Background] Schecter A, Colacino J, Haffner D, Patel K, Opel M, Papke O, Birnbaum L. Perfluorinated compounds, polychlorinated biphenyls, and organochlorine pesticide contamination in composite food samples from Dallas, Texas, USA. Environ Health Perspect. 2010 Jun;118(6):796-802. doi: 10.1289/ehp.0901347. Epub 2010 Feb 10. PMID 20146964
- [Background] Schecter A, Haffner D, Colacino J, Patel K, Papke O, Opel M, Birnbaum L. Polybrominated diphenyl ethers (PBDEs) and hexabromocyclodecane (HBCD) in composite U.S. food samples. Environ Health Perspect. 2010 Mar;118(3):357-62. doi: 10.1289/ehp.0901345. Epub 2009 Oct 28. PMID 20064778
- [Background] Lee DH, Steffes MW, Sjodin A, Jones RS, Needham LL, Jacobs DR Jr. Low dose of some persistent organic pollutants predicts type 2 diabetes: a nested case-control study. Environ Health Perspect. 2010 Sep;118(9):1235-42. doi: 10.1289/ehp.0901480. Epub 2010 May 5. PMID 20444671
- [Background] Lee DH, Lee IK, Jin SH, Steffes M, Jacobs DR Jr. Association between serum concentrations of persistent organic pollutants and insulin resistance among nondiabetic adults: results from the National Health and Nutrition Examination Survey 1999-2002. Diabetes Care. 2007 Mar;30(3):622-8. doi: 10.2337/dc06-2190. PMID 17327331
- [Background] Patterson DG Jr, Wong LY, Turner WE, Caudill SP, Dipietro ES, McClure PC, Cash TP, Osterloh JD, Pirkle JL, Sampson EJ, Needham LL. Levels in the U.S. population of those persistent organic pollutants (2003-2004) included in the Stockholm Convention or in other long range transboundary air pollution agreements. Environ Sci Technol. 2009 Feb 15;43(4):1211-8. doi: 10.1021/es801966w. PMID 19320182
- [Background] Smith D. Worldwide trends in DDT levels in human breast milk. Int J Epidemiol. 1999 Apr;28(2):179-88. doi: 10.1093/ije/28.2.179. PMID 10342677
- [Background] Centers for Disease Control and Prevention. Fourth National Report on Human Exposure to Environmental Chemicals. Atlanta, GA: Centers for Disease Control and Prevention; 2009. Available at: http://www.cdc.gov/exposurereport/pdf/FourthReport.pdf.
- [Background] Eskenazi B, Chevrier J, Rauch SA, Kogut K, Harley KG, Johnson C, Trujillo C, Sjodin A, Bradman A. In utero and childhood polybrominated diphenyl ether (PBDE) exposures and neurodevelopment in the CHAMACOS study. Environ Health Perspect. 2013 Feb;121(2):257-62. doi: 10.1289/ehp.1205597. Epub 2012 Nov 15. PMID 23154064
- [Background] Hsu MS, Hsu KY, Wang SM, Chou U, Chen SY, Huang NC, Liao CY, Yu TP, Ling YC. A total diet study to estimate PCDD/Fs and dioxin-like PCBs intake from food in Taiwan. Chemosphere. 2007 Apr;67(9):S65-70. doi: 10.1016/j.chemosphere.2006.05.116. Epub 2007 Jan 9. PMID 17215025
- [Background] Tsutsumi T, Yanagi T, Nakamura M, Kono Y, Uchibe H, Iida T, Hori T, Nakagawa R, Tobiishi K, Matsuda R, Sasaki K, Toyoda M. Update of daily intake of PCDDs, PCDFs, and dioxin-like PCBs from food in Japan. Chemosphere. 2001 Dec;45(8):1129-37. doi: 10.1016/s0045-6535(01)00151-5. PMID 11695626
- [Background] Li J, Zhang L, Wu Y, Liu Y, Zhou P, Wen S, Liu J, Zhao Y, Li X. A national survey of polychlorinated dioxins, furans (PCDD/Fs) and dioxin-like polychlorinated biphenyls (dl-PCBs) in human milk in China. Chemosphere. 2009 May;75(9):1236-42. doi: 10.1016/j.chemosphere.2009.01.073. Epub 2009 Feb 28. PMID 19251302
- [Background] Polder A, Thomsen C, Lindstrom G, Loken KB, Skaare JU. Levels and temporal trends of chlorinated pesticides, polychlorinated biphenyls and brominated flame retardants in individual human breast milk samples from Northern and Southern Norway. Chemosphere. 2008 Aug;73(1):14-23. doi: 10.1016/j.chemosphere.2008.06.002. Epub 2008 Jul 23. PMID 18653208
- [Background] Elobeid MA, Padilla MA, Brock DW, Ruden DM, Allison DB. Endocrine disruptors and obesity: an examination of selected persistent organic pollutants in the NHANES 1999-2002 data. Int J Environ Res Public Health. 2010 Jul;7(7):2988-3005. doi: 10.3390/ijerph7072988. Epub 2010 Jul 23. PMID 20717554
- [Background] Magliano DJ, Loh VHY, Harding JL, Botton J, Shaw JE. Persistent organic pollutants and diabetes: a review of the epidemiological evidence. Diabetes Metab. 2014 Feb;40(1):1-14. doi: 10.1016/j.diabet.2013.09.006. Epub 2013 Nov 18. PMID 24262435
- [Background] Ibrahim MM, Fjaere E, Lock EJ, Naville D, Amlund H, Meugnier E, Le Magueresse Battistoni B, Froyland L, Madsen L, Jessen N, Lund S, Vidal H, Ruzzin J. Chronic consumption of farmed salmon containing persistent organic pollutants causes insulin resistance and obesity in mice. PLoS One. 2011;6(9):e25170. doi: 10.1371/journal.pone.0025170. Epub 2011 Sep 23. PMID 21966444
- [Background] Ibrahim MM, Fjaere E, Lock EJ, Froyland L, Jessen N, Lund S, Vidal H, Ruzzin J. Metabolic impacts of high dietary exposure to persistent organic pollutants in mice. Toxicol Lett. 2012 Nov 23;215(1):8-15. doi: 10.1016/j.toxlet.2012.09.022. Epub 2012 Oct 4. PMID 23041606
- [Background] Remillard RB, Bunce NJ. Linking dioxins to diabetes: epidemiology and biologic plausibility. Environ Health Perspect. 2002 Sep;110(9):853-8. doi: 10.1289/ehp.02110853. PMID 12204817
- [Background] Lee DH, Steffes MW, Sjodin A, Jones RS, Needham LL, Jacobs DR Jr. Low dose organochlorine pesticides and polychlorinated biphenyls predict obesity, dyslipidemia, and insulin resistance among people free of diabetes. PLoS One. 2011 Jan 26;6(1):e15977. doi: 10.1371/journal.pone.0015977. PMID 21298090
- [Background] Tang M, Chen K, Yang F, Liu W. Exposure to organochlorine pollutants and type 2 diabetes: a systematic review and meta-analysis. PLoS One. 2014 Oct 15;9(10):e85556. doi: 10.1371/journal.pone.0085556. eCollection 2014. PMID 25329153
- [Background] Bloom MS, Jansing RL, Kannan K, Rej R, Fitzgerald EF. Thyroid hormones are associated with exposure to persistent organic pollutants in aging residents of upper Hudson River communities. Int J Hyg Environ Health. 2014 Apr-May;217(4-5):473-82. doi: 10.1016/j.ijheh.2013.09.003. Epub 2013 Sep 25. PMID 24138783
- [Background] Ribas-Fito N, Cardo E, Sala M, Eulalia de Muga M, Mazon C, Verdu A, Kogevinas M, Grimalt JO, Sunyer J. Breastfeeding, exposure to organochlorine compounds, and neurodevelopment in infants. Pediatrics. 2003 May;111(5 Pt 1):e580-5. doi: 10.1542/peds.111.5.e580. PMID 12728113
- [Background] Ribas-Fito N, Torrent M, Carrizo D, Munoz-Ortiz L, Julvez J, Grimalt JO, Sunyer J. In utero exposure to background concentrations of DDT and cognitive functioning among preschoolers. Am J Epidemiol. 2006 Nov 15;164(10):955-62. doi: 10.1093/aje/kwj299. Epub 2006 Sep 12. PMID 16968864
- [Background] Sagiv SK, Thurston SW, Bellinger DC, Tolbert PE, Altshul LM, Korrick SA. Prenatal organochlorine exposure and behaviors associated with attention deficit hyperactivity disorder in school-aged children. Am J Epidemiol. 2010 Mar 1;171(5):593-601. doi: 10.1093/aje/kwp427. Epub 2010 Jan 27. PMID 20106937
- [Background] Torres-Sanchez L, Schnaas L, Rothenberg SJ, Cebrian ME, Osorio-Valencia E, Hernandez Mdel C, Garcia-Hernandez RM, Lopez-Carrillo L. Prenatal p,p -DDE exposure and neurodevelopment among children 3.5-5 years of age. Environ Health Perspect. 2013 Feb;121(2):263-8. doi: 10.1289/ehp.1205034. Epub 2012 Nov 13. PMID 23151722
- [Background] Eskenazi B, Marks AR, Bradman A, Fenster L, Johnson C, Barr DB, Jewell NP. In utero exposure to dichlorodiphenyltrichloroethane (DDT) and dichlorodiphenyldichloroethylene (DDE) and neurodevelopment among young Mexican American children. Pediatrics. 2006 Jul;118(1):233-41. doi: 10.1542/peds.2005-3117. PMID 16818570
- [Background] Huang X, Lessner L, Carpenter DO. Exposure to persistent organic pollutants and hypertensive disease. Environ Res. 2006 Sep;102(1):101-6. doi: 10.1016/j.envres.2005.12.011. Epub 2006 Feb 3. PMID 16458884
- [Background] Sergeev AV, Carpenter DO. Exposure to Persistent Organic Pollutants Increases Hospitalization Rates for Myocardial Infarction with Comorbid Hypertension. Prim Prev Insights. 2010 Mar 23;2:1-9. doi: 10.4137/PPRI.S4332. PMID 21562627
- [Background] Lind L, Lind PM. Can persistent organic pollutants and plastic-associated chemicals cause cardiovascular disease? J Intern Med. 2012 Jun;271(6):537-53. doi: 10.1111/j.1365-2796.2012.02536.x. Epub 2012 Mar 30. PMID 22372998
- [Background] Lind PM, Penell J, Salihovic S, van Bavel B, Lind L. Circulating levels of p,p'-DDE are related to prevalent hypertension in the elderly. Environ Res. 2014 Feb;129:27-31. doi: 10.1016/j.envres.2013.12.003. Epub 2014 Jan 11. PMID 24528999
- [Background] Suarez-Lopez JR, Lee DH, Porta M, Steffes MW, Jacobs DR Jr. Persistent organic pollutants in young adults and changes in glucose related metabolism over a 23-year follow-up. Environ Res. 2015 Feb;137:485-94. doi: 10.1016/j.envres.2014.11.001. Epub 2015 Feb 23. PMID 25706918
- [Background] Schlummer M, Moser GA, McLachlan MS. Digestive tract absorption of PCDD/Fs, PCBs, and HCB in humans: mass balances and mechanistic considerations. Toxicol Appl Pharmacol. 1998 Sep;152(1):128-37. doi: 10.1006/taap.1998.8487. PMID 9772208
- [Background] Cohn WJ, Boylan JJ, Blanke RV, Fariss MW, Howell JR, Guzelian PS. Treatment of chlordecone (Kepone) toxicity with cholestyramine. Results of a controlled clinical trial. N Engl J Med. 1978 Feb 2;298(5):243-8. doi: 10.1056/NEJM197802022980504. PMID 74014
- [Background] Zeng E, ed. Persistent Organic Pollutants (POPs): Analytical Techniques, Environmental Fate and Biological Effects. Elsevier Science; 2015. Available at: https://books.google.com/books?id=YCAtBAAAQBAJ&pgis=1.
- [Background] Schecter A. Dioxins and Health Including Other Persistent Organic Pollutants and Endocrine Disruptors. John Wiley & Sons; 2012. Available at: https://books.google.com/books?id=4GI2sedIls4C&pgis=1
- [Background] Mochida Y, Fukata H, Matsuno Y, Mori C. Reduction of dioxins and polychlorinated biphenyls (PCBs) in human body. Fukuoka Igaku Zasshi. 2007 Apr;98(4):106-13. PMID 17533984
- [Background] Iida T, Nakagawa R, Hirakawa H, Matsueda T, Morita K, Hamamura K, Nakayama J, Hori Y, Guo YL, Chang FM, et al. Clinical trial of a combination of rice bran fiber and cholestyramine for promotion of fecal excretion of retained polychlorinated dibenzofuran and polychlorinated biphenyl in Yu-Cheng patients. Fukuoka Igaku Zasshi. 1995 May;86(5):226-33. PMID 7628813
- [Background] Jandacek RJ, Heubi JE, Buckley DD, Khoury JC, Turner WE, Sjodin A, Olson JR, Shelton C, Helms K, Bailey TD, Carter S, Tso P, Pavuk M. Reduction of the body burden of PCBs and DDE by dietary intervention in a randomized trial. J Nutr Biochem. 2014 Apr;25(4):483-8. doi: 10.1016/j.jnutbio.2014.01.002. Epub 2014 Jan 29. PMID 24629911
- [Background] Salas-Salvado J, Bullo M, Perez-Heras A, Ros E. Dietary fibre, nuts and cardiovascular diseases. Br J Nutr. 2006 Nov;96 Suppl 2:S46-51. doi: 10.1017/bjn20061863. PMID 17125533
- [Background] Ellis PR, Kendall CW, Ren Y, Parker C, Pacy JF, Waldron KW, Jenkins DJ. Role of cell walls in the bioaccessibility of lipids in almond seeds. Am J Clin Nutr. 2004 Sep;80(3):604-13. doi: 10.1093/ajcn/80.3.604. PMID 15321799
- [Background] Cassady BA, Hollis JH, Fulford AD, Considine RV, Mattes RD. Mastication of almonds: effects of lipid bioaccessibility, appetite, and hormone response. Am J Clin Nutr. 2009 Mar;89(3):794-800. doi: 10.3945/ajcn.2008.26669. Epub 2009 Jan 14. PMID 19144727
- [Background] Novotny JA, Gebauer SK, Baer DJ. Discrepancy between the Atwater factor predicted and empirically measured energy values of almonds in human diets. Am J Clin Nutr. 2012 Aug;96(2):296-301. doi: 10.3945/ajcn.112.035782. Epub 2012 Jul 3. PMID 22760558
- [Background] Vinson JA, Cai Y. Nuts, especially walnuts, have both antioxidant quantity and efficacy and exhibit significant potential health benefits. Food Funct. 2012 Feb;3(2):134-40. doi: 10.1039/c2fo10152a. Epub 2011 Dec 21. PMID 22187094
- [Background] Hennig B, Ormsbee L, McClain CJ, Watkins BA, Blumberg B, Bachas LG, Sanderson W, Thompson C, Suk WA. Nutrition can modulate the toxicity of environmental pollutants: implications in risk assessment and human health. Environ Health Perspect. 2012 Jun;120(6):771-4. doi: 10.1289/ehp.1104712. Epub 2012 Feb 22. PMID 22357258
- [Background] Lee DH, Porta M, Jacobs DR Jr, Vandenberg LN. Chlorinated persistent organic pollutants, obesity, and type 2 diabetes. Endocr Rev. 2014 Aug;35(4):557-601. doi: 10.1210/er.2013-1084. Epub 2014 Jan 31. PMID 24483949
- [Background] Lee DH, Lee IK, Song K, Steffes M, Toscano W, Baker BA, Jacobs DR Jr. A strong dose-response relation between serum concentrations of persistent organic pollutants and diabetes: results from the National Health and Examination Survey 1999-2002. Diabetes Care. 2006 Jul;29(7):1638-44. doi: 10.2337/dc06-0543. PMID 16801591
- [Background] Lee DH, Lind PM, Jacobs DR Jr, Salihovic S, van Bavel B, Lind L. Polychlorinated biphenyls and organochlorine pesticides in plasma predict development of type 2 diabetes in the elderly: the prospective investigation of the vasculature in Uppsala Seniors (PIVUS) study. Diabetes Care. 2011 Aug;34(8):1778-84. doi: 10.2337/dc10-2116. Epub 2011 Jun 23. PMID 21700918
- [Background] Zota AR, Park JS, Wang Y, Petreas M, Zoeller RT, Woodruff TJ. Polybrominated diphenyl ethers, hydroxylated polybrominated diphenyl ethers, and measures of thyroid function in second trimester pregnant women in California. Environ Sci Technol. 2011 Sep 15;45(18):7896-905. doi: 10.1021/es200422b. Epub 2011 Aug 19. PMID 21830753
- [Background] Clinical and Laboratory Standards Institute. Procedures for the Collection of Diagnostic Blood Specimens by Venipuncture: Approved Standard. Sixth. (Ernst D, ed.). Wayne, Pa.: Clinical and Laboratory Standards Institute; 2007.
- [Background] Hoh E, Lehotay SJ, Mastovska K, Ngo HL, Vetter W, Pangallo KC, Reddy CM. Capabilities of direct sample introduction--comprehensive two-dimensional gas chromatography--time-of-flight mass spectrometry to analyze organic chemicals of interest in fish oils. Environ Sci Technol. 2009 May 1;43(9):3240-7. doi: 10.1021/es803486x. PMID 19534141
- [Background] Hoh E, Dodder NG, Lehotay SJ, Pangallo KC, Reddy CM, Maruya KA. Nontargeted comprehensive two-dimensional gas chromatography/time-of-flight mass spectrometry method and software for inventorying persistent and bioaccumulative contaminants in marine environments. Environ Sci Technol. 2012 Aug 7;46(15):8001-8. doi: 10.1021/es301139q. Epub 2012 Jul 9. PMID 22712571
- [Background] Hoh E, Lehotay SJ, Pangallo KC, Mastovska K, Ngo HL, Reddy CM, Vetter W. Simultaneous quantitation of multiple classes of organohalogen compounds in fish oils with direct sample introduction comprehensive two-dimensional gas chromatography and time-of-flight mass spectrometry. J Agric Food Chem. 2009 Apr 8;57(7):2653-60. doi: 10.1021/jf900462p. PMID 19265383
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ. 2001 Nov 10;323(7321):1123-4. doi: 10.1136/bmj.323.7321.1123. No abstract available. PMID 11701584
- [Background] Mattes RD, Kris-Etherton PM, Foster GD. Impact of peanuts and tree nuts on body weight and healthy weight loss in adults. J Nutr. 2008 Sep;138(9):1741S-1745S. doi: 10.1093/jn/138.9.1741S. PMID 18716179
- [Background] Baer DJ, Gebauer SK, Novotny JA. Walnuts Consumed by Healthy Adults Provide Less Available Energy than Predicted by the Atwater Factors. J Nutr. 2016 Jan;146(1):9-13. doi: 10.3945/jn.115.217372. Epub 2015 Nov 18. PMID 26581681